CLINICAL TRIAL: NCT01244256
Title: Isolation and Comparative Efficacy of the Combination of beclometasona0, 025% + Gentamicin 0.1% + Clotrimazole 1% Topical Dermatological Cream of GLENMARK PHARMACEUTICALS, in Patients Infected With Acne
Brief Title: Efficacy and Comparative of the Association Beclomethasone Clotrimzaol + Gentamicin in Patients With Acne Contaminated
Acronym: acne
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Responsible Party: Principal Investigator, Azidus Brasil, Principal Investigator Dr. Alexandre Frederico, Azidus Brasil
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BCGGLE10407
Record Dates: First submitted 2010-10-22; First posted 2010-11-19 (Estimated); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Folliculitis
MeSH Terms: conditions — Folliculitis | interventions — Clotrimazole; Gentamicins; Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment with Clotrimazole + Gentamicin + Beclomethasone (Experimental)
  Interventions: Drug: Clotrimazole + Gentamicin + Beclomethasone
- Treatment with Clotrimazole + Gentamicin (Active Comparator)
  Interventions: Drug: Clotrimazole + Gentamicin

INTERVENTIONS:
Drug: Clotrimazole + Gentamicin + Beclomethasone — Treatment with Clotrimazole + Gentamicin + Beclomethasone
  Arms: Treatment with Clotrimazole + Gentamicin + Beclomethasone
Drug: Clotrimazole + Gentamicin — Treatment with Clotrimazole + Gentamicin
  Arms: Treatment with Clotrimazole + Gentamicin

SUMMARY:
The objective of this trial is to evaluate the comparative efficacy of the combination of Clotrimazole + Gentamicin + Beclomethasone in study subjects with a condition of contaminated dermatosis showing bilateral symmetrical lesions.

DETAILED DESCRIPTION:
The specific objective is to evaluate, by means of analytical propedeutics medical improvement in clinical signs and symptoms related to acne infected, the use of the association: Clotrimazole, Gentamicin and Beclomethasone versus association: Clotrimazole and Gentamicin, which will first be randomized.

The study should be conducted with 20 research subjects aged over 18 years, of both sexes, showing the framework of bilateral lesions infected with acne, at any stage of evolution. The study subjects will receive treatment with both products, so they can use one in each lesion chosen at random, double-blind.

Thus, the proven efficacy and safety and taking all possible adverse events reported, the study sponsor hopes to obtain registration with the Ministry of Health of this new association in the country.

The association made a proposal was developed by the Laboratory Glenmark Pharmaceuticals Ltd..

ELIGIBILITY:
Inclusion Criteria:

* Subject search of both sexes, regardless of color or social class
* From age to 18, with good mental health
* Carriers of two outbreaks of acne contaminated
* Subjects who agree to return follow-up visits
* Research subjects who agree to participate and sign the Deed of Consent

Exclusion Criteria:

* Subject Research carriers of susceptibility to gentamicin
* Research subjects suffering from sensitivity to clotrimazole
* Research subjects suffering from sensitivity to beclomethasone
* Research subjects who are making use of steroids or steroidal anti-inflammatory and non-steroidal drugs or who made use of topical or oral 15 days ago
* Research subjects who are doing immunosuppressive treatment
* Research subjects with a diagnosis of eosinophilic folliculitis or Pseudo-folliculitis barbae and groin
* Pregnant and lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-04 (Actual); Primary Completion 2007-08 (Actual); Study Completion 2007-09

PRIMARY OUTCOMES:
Efficacy of the treatment in patient with infected dermatoses | 21 days of treatment

SECONDARY OUTCOMES:
evaluate the safety and tolerability of both formulations in the course of treatmen | 21 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Frederico, médico, Principal Investigator — Azidus Brasil
Locations (1):
- LAL Clinica, Valinhos, São Paulo, Brazil